CLINICAL TRIAL: NCT01586182
Title: Stereotactic Boost for Poor-Prognosis Oropharyngeal Squamous Cell Carcinoma
Brief Title: Stereotactic Boost for Oropharyngeal Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Local IRB closed the study due to poor accural.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Roy B. Tishler, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-037
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
Keywords: poor prognosis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Boost (Experimental): Escalating doses of stereotactic body radiation therapy (SBRT)
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Starting dose is 5.5 Gy x 2 boosts in addition to 57.24 Gy to the primary disease

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational intervention (in this case, the stereotactic radiation boost). Phase I studies also try to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the stereotactic radiation treatment is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved a stereotactic radiation boost for your type of cancer.

In this research study, the investigators are looking for the highest dose of the stereotactic radiation boost that can be given safely. Because the stereotactic radiation boost is so precise, the investigators are testing whether it can be used to increase the dose to the primary tumor without significantly increasing the side effects you experience; the goal is to improve the likelihood of successfully treating the tumor.

DETAILED DESCRIPTION:
After confirming that you are eligible for this study and your willingness to participate in it, we will perform a radiation treatment stimulation, or "mapping session," within the next two weeks. You may or may not receive intravenous contrast during the process, which allows your physician to better see the blood vessels in your neck. You will be placed in a mask during this process to help keep you in the same place during each treatment. All of this is part of standard radiation treatment.

Approximately 14 days later, you will start radiation treatment to your primary tumor site and to your lymph nodes and chemotherapy in the same week. The chemotherapy will continue to be given one time per week during each week of treatment. You will receive radiation treatment 5 days a week for seven weeks. One day each during the first and second weeks of treatment, instead of the typical radiation dose, you will receive a dose of the stereotactic radiation boost to the site of the primary tumor (total of 2 doses of stereotactic radiotherapy).

Because we are looking for the highest dose of the stereotactic radiation boost that can be administered safely without severe or unmanageable side effects, not everyone who participates in this research study will receive the same dose of the stereotactic radiation boost. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses. We are testing 3 different dose levels for the stereotactic radiation boost; your dose will be one of those 3 doses.

The chemotherapy will be given one time per week, each week, for the duration of the radiation treatment (7 weeks). The chemotherapy is delivered through intravenous fluids that run through a vein in your arm. This is the same chemotherapy that you would receive if you were not participating in the study.

You will be seen by your radiation oncologist at least once every week during treatment.

After the final dose of radiation treatment all subsequent follow-up visits and tests are performed in accordance with standard cancer care. You will see your radiation oncologist, with or without the medical oncologist, at the following time intervals: 1 week after treatment ends, 1 month after treatment ends, 2 months after treatment ends, and then every 3 months for two years. You will undergo a PET-CT scan and neck CT scan at the time of the 3 month appointment.

You will be on the study treatment for about 7 weeks and your progress will be followed as part of the study for 2 years after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated histologically or cytologically confirmed T2-4, N0-3 HPV16-negative oropharyngeal squamous cell carcinoma or HPV16 positivity with at least a 10 pack-year smoking habit
* Measurable disease
* Life expectancy of greater than 6 months

Exclusion Criteria:

* Other active malignancy within the past 5 years (except for non-melanoma skin cancer or carcinoma in situ of the cervix)
* Primary tumor size > 6 cm
* Prior history of head and neck radiotherapy
* Receiving any other study agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding
* HIV positive on combination antiretroviral therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Determination of MTD | 2 years
  Determination of the MTD and dose-limiting toxicities of a stereotactic boost to chemoradiotherapy for poor-prognosis oropharyngeal squamous cell carcinoma
Two Year Local Control Rate | 2 years
  Local failure is defined as biopsy-proven recurrent disease

SECONDARY OUTCOMES:
Safety and Tolerability of Stereotactic Boost | 2 years
  To evaluate the safety and tolerability of a stereotactic boost to chemoradiotherapy, including both acute and long-term toxicity
Overall Survival | 2 years
  To determine the 2 year overall survivial
Disease-Free Survival | 2 years
  To determine the 2-year disease-free survival

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts